CLINICAL TRIAL: NCT01571843
Title: Effect of Mechanical Loading on Radius Bone Density and Microarchitecture in Primary Hyperparathyroidism
Brief Title: Radius Loading in Primary Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John P. Bilezikian, Dorothy L. and Daniel H. Silberberg Professor of Medicine and Pharmacology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAE6548; R01DK032333 (NIH)
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Primary Hyperparathyroidism; Bone Diseases, Metabolic; Osteoporosis, Postmenopausal; Bone Loss, Postmenopausal
Keywords: Hyperparathyroidism, Primary; Bone Diseases, Metabolic; Osteoporosis, Postmenopausal; Bone Loss, Postmenopausal
MeSH Terms: conditions — Hyperparathyroidism, Primary; Bone Diseases, Metabolic; Osteoporosis, Postmenopausal | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PHPT/ Walking + Forearm exercise (Experimental): Ten participants with PHPT will be randomized to the intervention of 52 weeks of the forearm exercise program plus walking.
  Interventions: Other: Forearm exercise program
- PHPT/ Walking alone (Placebo Comparator): Ten participants with PHPT will be randomized to the intervention of 52 weeks of the walking program alone. Walking will consist of 30 minutes at a moderate pace every other day for 52 weeks.
  Interventions: Other: Walking program
- Osteopenia/ Walking + Forearm exercise (Active Comparator): Ten healthy, postmenopausal women with osteopenia will be randomized to the intervention of 52 weeks of the forearm exercise program plus walking.
  Interventions: Other: Forearm exercise program
- Osteopenia/ Walking alone (Placebo Comparator): Ten healthy, postmenopausal women with osteopenia will be randomized to the intervention of 52 weeks of the walking program alone. Walking will consist of 30 minutes at a moderate pace every other day for 52 weeks.
  Interventions: Other: Walking program

INTERVENTIONS:
Other: Forearm exercise program — Participants assigned to forearm exercise will receive training in forearm strengthening exercises from a doctoral occupational therapy student. Participants will be taught 8 exercises and are performed at home. The exercise program is designed to take about 30 minutes per session.
  Other Names: Mechanical Loading
  Arms: Osteopenia/ Walking + Forearm exercise; PHPT/ Walking + Forearm exercise
Other: Walking program — Walking will consist of 30 minutes at a moderate pace every other day for 52 weeks. The walking program for all participants constitutes the control/placebo comparator.
  Other Names: Walking
  Arms: Osteopenia/ Walking alone; PHPT/ Walking alone

SUMMARY:
The purpose of the study is to determine the effect of forearm exercise on forearm bone density in post-menopausal women with or without primary hyperparathyroidism.

The investigators hypothesize that forearm exercise will increase forearm bone density in patients with primary hyperparathyroidism more so than in patients without primary hyperparathyroidism.

DETAILED DESCRIPTION:
Primary hyperparathyroidism (PHPT), a disease characterized by excess parathyroid hormone (PTH) and high blood calcium, is one of the most common endocrine disorders.

PHPT is seen most often in post-menopausal women. Kidney stones and bone deformities were prominent manifestations of the disease in the past, however, PHPT is now primarily asymptomatic due to incidental detection of high blood calcium levels.

Many patients with PHPT, however, have low bone mineral density (BMD) when bone mass is measured by dual energy x-ray absorptiometry (DXA), primarily at the forearm.

There is no effective medical therapy which increases bone density at the forearm in patients with PHPT. PTH both builds and breaks down bone, and the pathways by which PTH mediates these actions are beginning to be identified. Prior research suggests that mechanical loading shifts PTH towards building bone. Arm exercise is an attractive option for the treatment of low forearm BMD in patients with PHPT since it is often the site most affected by excess PTH.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for primary hyperparathyroidism group:

1. Primary hyperparathyroidism (defined by an elevated serum calcium and concomitantly elevated or inappropriately normal PTH)
2. Female sex, postmenopausal status for at least five years, ages 45-80
3. English- or Spanish-speaking
4. DXA T-score less than -1.0 at the one-third radius
5. Physically capable of exercise
6. 25-hydroxyvitamin D >20 ng/mL. The latter inclusion criterion will lead to the enrollment of some individuals whose vitamin D stores will not be frankly low. We feel, however, that it is better to study subjects in their usual state rather than replacing them with vitamin D which could add another variable that would further complicate this pilot study.

Inclusion criteria for the osteopenic control:

1. Female sex, postmenopausal status for at least five years ages 45-80
2. English- or Spanish-speaking
3. DXA T-score less than -1.0 at the one-third radius
4. Physically capable of exercise
5. Normal serum calcium and PTH level
6. 25-hydroxyvitamin D >20 ng/mL

Exclusion Criteria:

1. Men, premenopausal women, women less than age 45 or greater than age 80
2. Familial hypocalciuric hypercalcemia
3. Current or prior use of bisphosphonates (alendronate or risedronate (within 12 months), ibandronate (within 6 months), other bisphosphonate (2 years)
4. Current use of cinacalcet
5. Current or prior use of estrogen replacement therapy (within 2 years)
6. Planned parathyroidectomy (within one year)
7. Planned initiation of bisphosphonates
8. DXA T-score greater than -1.0 at the one-third radius
9. Cardiovascular disease or uncontrolled hypertension
10. Exercise-limiting pulmonary diseases
11. Malignancy other than non-melanomatous skin cancer or microscopic thyroid cancer (within 5 years)
12. Renal failure
13. Secondary hyperparathyroidism
14. Celiac disease
15. Physical/orthopedic disabilities and neurologic disorders or vasculopathies that would place the subjects at risk or limit their ability to perform exercise (eg. arthritis, carpal tunnel syndrome, rotator cuff injury, etc)
16. Moderate or high physical activity (category 2 or 3) as assessed by the IPAQ questionnaire. This latter exclusion criterion is a measure of baseline physical activity and looks to exclude those who would have a lower likelihood of benefit by baseline participation in an exercise program.
17. Protected individuals (institutionalized), prisoners, and any other prospective participant who might not be able to give voluntary informed consent.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with improved bone mass and bone quality at the 1/3 radius | 1 year
  The primary outcome is proportion of subjects with improved bone mass and bone quality at the 1/3 radius over one year.

CONTACTS AND LOCATIONS:
Overall Officials: John P Bilezikian, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- See also: Click here for more information about this study, "The Effect of Mechanical Loading on Radius Bone Density and Microarchitecture in Primary Hyperparathyroidism" — http://www.columbiamedicine.org/divisions/Endo/index.shtml